CLINICAL TRIAL: NCT03565484
Title: 14-Day Antimicrobial Susceptibility Testing Guided Therapy Versus Personal Medication History Guided Therapy as a Rescue Treatment of Helicobacter Pylori Infection-A Randomized Controlled Trail
Brief Title: Antimicrobial Susceptibility Testing Guided Therapy Versus Empirical Therapy for the Rescue Treatment of Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017SDU-QILU-G004
Record Dates: First submitted 2018-06-18; First posted 2018-06-21 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Antimicrobial Susceptibility Testing; Rescue Therapy
MeSH Terms: interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Antimicrobial susceptibility testing guided therapy (Experimental): 14d bismuth quadruple therapy based on susceptibility test.
  Interventions: Drug: susceptibility guided therapy
- Personal medication history guided therapy (Experimental): 14d bismuth quadruple therapy based on previous medication history.
  Interventions: Drug: personal medication history guided therapy
- Salvage therapy for negative culture (Other): 14d bismuth quadruple therapy based on previous medication history.
  Interventions: Drug: personal medication history guided therapy
- Salvage therapy for failed eradication (Other): 14d bismuth quadruple therapy for salvage treatment.
  Interventions: Drug: salvage treatment for failed eradication

INTERVENTIONS:
Drug: susceptibility guided therapy — Patients will take a gastroscopy and 2 biopsies will be attained from antrum and gastric body for H.pylori culture and antimicrobial susceptibility testing (AST). The susceptibility of amoxicillin, clarithromycin, metronidazole, levofloxacin, furazolidone and tetracycline will be tested.Then patients with positive culture will be treated with a 14-day quadruple therapy for the H.pylori eradication. The regimen contains rabeprazole 20mg bid, colloidal bismuth pectin 200mg bid, and two sensitive antibiotics determined by AST. Dose of two sensitive antibiotics are listed as follows : amoxicillin 1000mg bid, clarithromycin 500mg bid, tinidazole 500mg tid, levofloxacin 500mg qd, furazolidone 100mg bid, tetracycline 500mg qid.
  Arms: Antimicrobial susceptibility testing guided therapy
Drug: personal medication history guided therapy — Patients will be treated with a 14-day emprical tailored quadruple therapy for the H.pylori eradication. The regimen contains rabeprazole 20mg bid， colloidal bismuth pectin 200mg bid and two antibiotics based on personal medication history. If the patient doesn't have levofloxacin history, he will be treated with amoxicillin 1000mg bid plus levofloxacin 500mg bid. Otherwise, he will be treated with amoxicillin 1000mg bid and furazolidone 100mg bid.
  Arms: Personal medication history guided therapy; Salvage therapy for negative culture
Drug: salvage treatment for failed eradication — If the patients failed with AST guided eradication therapy or empirical therapy, patients will be treated with another 14-day bismuth-based quadruple therapy. The regimen contains rabeprazole 20mg bid, colloidal bismuth pectin 200mg bid, tetracycline 500mg qid and furazolidone 100mg bid.
  Arms: Salvage therapy for failed eradication

SUMMARY:
The purpose of this study is to assess efficacy of 14-day antimicrobial susceptibility test guided quadruple therapy for the rescue treatment of Helicobacter pylori infection, then comparing it with 14-day personal medication history guided therapy to tell which one has a better performance in both efficacy and safety.

DETAILED DESCRIPTION:
Helicobacter pylori (H.pylori), which infects about 50% of the global population, has been recognized as a main risk factor of multiple gastric pathology, especially non-cardiac gastric cancer. Strong evidence supports that H.pylori eradication is an effective approach to reduce the incidence of those pathological processes. Antimicrobial susceptibility test can pick out sensitive drugs to kill Helicobacter pylori, and reduce secondary drug resistance. But, there is a lack of high quality RCT to compare its efficacy with empirical regimen in the rescue treatment.

This study aims to assess the efficacy of 14-day antimicrobial susceptibility test guided quadruple therapy for the rescue treatment of Helicobacter pylori infection. Comparing this regimen with 14-day personal Medication History guided therapy to tell which one is better in clinic practice. Alterations in H.pylori assosicated dyspepsia and safety outcomes will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-70 with H. pylori infection. Patients with previous H. pylori eradication therapy for one or two times.

Exclusion Criteria:

Patients unable or unwilling to receive gastroscopy; Patients treated with H2-receptor antagonist, PPI, bismuth and antibiotics in the previous 4 weeks; Patients with gastrectomy, acute GI bleeding and advanced gastric cancer; Patients with known or suspected allergy to study medications; Currently pregnant or lactating; Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rates in 2 groups | 6 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients. The PP analysis is limited to patients who take over 80% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
The rate of improving dyspepsia symptoms after Helicobacter pylori eradication. | 6 months
  Dyspepsia symptoms will be measured using a 8-point Likert scale, and patients rate their symptoms from 0 (none) to 8 (severe) before and after the Helicobacter pylori eradication.

OTHER OUTCOMES:
The rate of adverse events happening | 6 months
  Similarly, adverse events will also be measured by the Likert scale.
The rate of good compliance | 6 months
  Patients taken over 80% of drugs are considered to have a good compliance.
Difference of cost per patient for each eradication achieved in two groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China